CLINICAL TRIAL: NCT05410925
Title: Efficacy and Safety of a Half-dose Bolus of r-SAK Prior to Primary PCI in ST-elevation Myocardial Infarction: a Multicenter Randomized Double-blind Placebo-controlled Trial (OPTIMA-6)
Brief Title: Efficacy and Safety of a Half-dose Bolus of r-SAK Prior to Primary PCI in ST-elevation Myocardial Infarction
Acronym: OPTIMA-6
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Director of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 018
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST Elevation Myocardial Infarction; Recombinant Staphylokinase; Thrombolysis
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- r-SAK group (Experimental): intravenous injection of single-bolus 5 mg r-SAK in 3 min
  Interventions: Drug: Recombinant staphylokinase
- placebo group (Placebo Comparator): intravenous injection of placebo in 3 min
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant staphylokinase — Intravenous injection of r-SAK is administered within 10 minutes after diagnosis of acute ST-segment elevation myocardial infarction
  Arms: r-SAK group
Drug: Placebo — Intravenous injection of placebo is administered within 10 minutes after diagnosis of acute ST-segment elevation myocardial infarction
  Arms: placebo group

SUMMARY:
As an effective treatment for acute ST-segment elevation myocardial infarction (STEMI), early reperfusion may reduce the infarct size and improve the prognosis of patients. However, it remains uncertain whether adjunctive thrombolytic therapy administered immediately prior to primary percutaneous coronary intervention (PCI) improves outcomes in patients undergoing the procedure within 120 minutes.

In this investigator-initiated, prospective, multi-center, randomized, double-blind, placebo-controlled trial, subjects meeting the inclusion/exclusion criteria should be randomly assigned 1:1 to the trial group (r-SAK) or the control group (placebo). The risk of major adverse cardiovascular events within 90 days will be observed.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is a serious and critical disease that causes acute coronary artery stenosis, spasm or occlusion due to the rupture or erosion of coronary artery plaque, resulting in myocardial ischemia and necrosis. Myocardial ischemia and necrosis can cause myocardial cell loss, ventricular remodeling and local inflammatory reaction, leading to decreased cardiac output or increased intracardiac pressure, and eventually progress to heart failure (HF), which seriously affects the prognosis of patients. The FAST-MI study found that 37.5% of AMI patients were complicated with HF, and the 1-year mortality of these patients was significantly increased. Early reperfusion treatment as an effective means of AMI treatment can promote myocardial reperfusion, save dying myocardium and reduce infarct area, which is of great significance to improve the clinical prognosis of patients.

At this stage, many primary hospitals do not have the conditions for emergency percutaneous coronary intervention (PCI). Transferring patients to PCI hospitals takes a lot of time, delaying the best time for early reperfusion treatment. In addition, the thrombus burden in the coronary artery increases with the prolongation of ischemia time. Stent implantation in the coronary artery with excessive thrombus burden is prone to slow blood flow or no reflow, resulting in the occurrence of major adverse cardiovascular events (MACE). In view of the above problems, guidelines suggest that if the estimated transit time is more than 120 minutes, thrombolytic therapy should be performed before transport; If the estimated transfer time is less than 120 minutes, it can be directly transferred to the PCI hospital.

However, it remains uncertain whether adjunctive thrombolytic therapy administered immediately prior to primary PCI improves outcomes in patients undergoing the procedure within 120 minutes ("facilitated PCI"). Multiple previous studies comparing facilitated PCI with primary PCI found facilitated PCI to be inferior in terms of clinical outcomes, while other studies based on reduced-dose thrombolysis confirmed the superiority of facilitated PCI in better patency of infarct-related artery (IRA). Recombinant staphylokinase (r-SAK), as the third-generation thrombolytic agent, may serve as the potential thrombolytic drug to contemporary facilitated PCI by virtue of its high fibrinolytic activity and fibrin selectivity.

Staphylokinase (SAK) is produced by Staphylococcus aureus and it is a protein containing 136 amino acid residues. Its ability for dissolving blood clots was first discovered in 1948. Studies have shown that SAK is not directly convert plasminogen (PLG) into plasminogen (PLi), but first combines with PLG in a 1:1 ratio to form a complex. The complex can lead to the exposure of PLG active site, from single chain to double chain PLi, resulting to form an active SAK-PLI complex, which subsequently activates PLG molecules. Then PLG transforms into PLi and further dissolve the thrombus.

R-SAK was developed in 1990 by Shanghai Institute of Plant and Biological Physiology. It is a gene recombinant drug prepared by molecular cloning of SAK gene in Escherichia coli. Its biological characteristics are very similar to natural SAK, and r-SAK is a highly fibrin-specific fibrinolysis agent. R-SAK is considered to be one of the most promising thrombolytic drugs due to its high thrombolysis activity (especially in platelet-rich arterial thrombosis), inactivation of system fibrinolysis, and few side effects. Clinical studies have shown that the efficacy of r-SAK in the treatment of AMI is better than urokinase, comparable to RT-PA, and it does not increase serious bleeding complications such as intracranial hemorrhage.

In terms of pharmacokinetics, r-SAK has a fast distribution and a long action time in human body. Half-lives of distribution term is 13.30±2.06min and elimination term is 67.94±21.39min when intravenous injection 10 mg r-SAK in 30min. A single bolus of r-SAK as early as possible during the first medical contact (such as prehospital care or primary hospitals or medical centers with conditional PCI) can maximize the time window for reperfusion therapy.

Achieving early reperfusion by means of facilitated PCI is consistent with the core of STEMI treatment, but the efficacy and safety of facilitated PCI are still controversial. OPTIMA-6, designed as shorter symptom onset to treatment time, a half-dose thrombolytic agent, and upstream use of the potent antiplatelet agent, will therefore evaluate the efficacy and safety of a half-dose bolus of r-SAK vs. placebo prior to primary PCI to inform clinical practice of contemporary facilitated PCI in patients with STEMI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, weight ≥45 kg
2. Diagnosed as STEMI (meeting the following two conditions simultaneously)

   1. Ischemic chest pain lasts ≥ 30 minutes
   2. ECG indicates that ST-segment elevation of two or more contiguous precordial leads ≥ 0.1 mV, or ST-segment elevation of two or more contiguous precordial leads ≥ 0.2 mV
3. Time from onset of persistent chest pain to randomization ≤12 hours
4. Primary PCI expected to be performed ≥30 minutes, and ≤120 minutes

Exclusion Criteria:

1. Cardiogenic shock
2. Active bleeding or known at high risk of bleeding (including grade Ⅲ or Ⅳ retinopathy or retinal gastrointestinal or urinary tract hemorrhage within the past 1 month)
3. Ischemic stroke or TIA in the past 6 months
4. History of hemorrhagic stroke
5. Known intracranial aneurysm
6. Severe trauma, surgery or head injury within 1 month
7. Suspected aortic dissection or infective endocarditis
8. Puncture with difficult hemostasis by compression within 1 month (e.g., visceral biopsy, compartment puncture)
9. Currently taking anticoagulants
10. Poorly controlled hypertension ( ≥180/110 mmHg)
11. Severe hepatic or renal impairment indicated by the consultation or previous history (glutamic-pyruvic transaminase or glutamic oxalacetic transaminase >3 times upper limit of normal value; eGFR <15 ml/min/1.73m^2, calculated based on CKD-EPI)
12. Known allergy to r-SAK
13. Pregnancy, lactation, or planning for pregnancy
14. History of chronic total occlusion, myocardial infarction or CABG
15. Having taken antiplatelet drugs other than aspirin and ticagrelor, such as clopidogrel, prasugrel or cilostazol after the symptom onset
16. Patients with other conditions that made them unsuitable to be recruited at the discretion of the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2260 (Estimated)
Dates: Start 2023-04-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
MACE | Within 90 days
  Defined as a composite of all-cause death, reinfarction, unplanned target vessel revascularization, heart failure or cardiogenic shock, major ventricular arrhythmia

SECONDARY OUTCOMES:
Each of the following cardiac and cerebrovascular events | Within 90 days
  Including all-cause death, cardiovascular death, reinfarction, stroke, unplanned target vessel revascularization, heart failure or cardiogenic shock, major ventricular arrhythmia, cardiogenic rehospitalization, ventricular septal rupture, papillary muscle rupture, cardiac rupture, ventricular aneurysm
NT-proBNP | 1 day before discharge or day 7, day 90±3
  The level of NT-proBNP
CMR indexes | Day 5
  Including infarct size, left ventricular ejection fraction (LVEF), microvascular obstruction (MVO) and intramuscular hemorrhage (IMH), assessed by cardiac magnetic resonance (CMR)
LVEF assessed by echocardiogram | Day 90±3
  LVEF assessed by echocardiogram
The percentage of TIMI flow grade 2 and 3 prior to PCI | Immediately prior to PCI
  The percentage of thrombolysis in myocardial infarction (TIMI) flow grade 2 and 3 prior to PCI
The percentage of TIMI flow grade 3 prior to PCI | Immediately prior to PCI
  The percentage of TIMI flow grade 3 prior to PCI
The percentage of TIMI flow grade 2 and 3 after PCI | Immediately after PCI
  The percentage of TIMI flow grade 2 and 3 after PCI
The percentage of TIMI flow grade 3 after PCI | Immediately after PCI
  The percentage of TIMI flow grade 3 after PCI
MACE | Within 360 days
  Defined as a composite of all-cause death, reinfarction, unplanned target vessel revascularization, heart failure or cardiogenic shock, major ventricular arrhythmia
Each of the following cardiac and cerebrovascular events | Within 360 days
  Including all-cause death, cardiovascular death, reinfarction, ischemic stroke, unplanned target vessel revascularization, heart failure or cardiogenic shock, major ventricular arrhythmia, cardiogenic rehospitalization, ventricular septal rupture, papillary muscle rupture, cardiac rupture, ventricular aneurysm
NT-proBNP | Day 360±7
  The level of NT-proBNP
LVEF assessed by echocardiogram | Day 360±7
  LVEF assessed by echocardiogram

OTHER OUTCOMES:
Major bleeding events during hospitalization or within 7 days (BARC 3, 5) | During hospitalization or within 7 days
  Major bleeding events during hospitalization or within 7 days (BARC 3, 5)
Minor bleeding events during hospitalization or within 7 days (BARC 2) | During hospitalization or within 7 days
  Minor bleeding events during hospitalization or within 7 days (BARC 2)
Major bleeding events within 90 days (BARC 3, 5) | Within 90 days
  Major bleeding events within 90 days (BARC 3, 5)
Minor bleeding events within 90 days (BARC 2) | Within 90 days
  Minor bleeding events within 90 days (BARC 2)

CONTACTS AND LOCATIONS:
Overall Officials: Chunjian Li, PHD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (61):
- China (61):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Changzhou Second People's Hospital, Changzhou
  - Changzhou Wujin People's Hospital, Changzhou
  - The First People's Hospital of Changzhou, Changzhou
  - Chongqing Hospital of Jiangsu Province Hospital, Chongqing
  - The second Affiliated Hospital of Dalian Medical University, Dalian
  - Daqing Oilfield General Hospital, Daqing
  - Dongguan People's Hospital, Dongguan
  - Fengcheng People's Hospital, Fengcheng
  - General Hospital of Southern Theatre Command, Guangzhou
  - The Second Affiliated Hospital of Hainan Medical University, Hainan
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huai'an First People's Hospital, Huai'an
  - Huai'an Second People's Hospital, Huai'an
  - Donghai Country People's Hospital, Lianyungang
  - The First People's Hospital of Lianyungang, Lianyungang
  - The Second People's Hospital of Lianyungang, Lianyungang
  - Liyang Hospital of Jiangsu Province Hospital, Liyang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Tongren Hospital, Nanjing
  - Sir Run Run Hospital Nanjing Medical University, Nanjing
  - The Fourth Affiliated Hospital of Nanjing Medical University, Nanjing
  - Nanjing Qixia District Hospital, Nanning
  - Affiliated Hospital of Nantong University, Nantong
  - Nantong First People's Hospital, Nantong
  - The People's Hospital of Zhalaite, Neimeng
  - Qingdao Municipal Hospital, Qingdao
  - Qilu Hospital of Shandong University, Shandong
  - Renji Hospital affiliated to Shanghai Jiaotong University, Shanghai
  - Songjiang Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - The People's Hospital of Liaoning Province, Shenyang
  - Shenzhen People's Hospital, Shenzhen
  - Suining County People's Hospital, Suining
  - Nanjing Drum Tower Hospital Group Suqian Hospital, Suqian
  - Suqian First Hospital, Suqian
  - Suzhou Dushu Lake Hospital, Suzhou
  - Suzhou Municipal Hospital of Anhui Province, Suzhou
  - Suzhou Municipal Hospital, Suzhou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Wanbei Coal-Electricity Group General Hospital, Suzhou
  - Taihe County Traditional Chinese Medicine Hospital, Taihe
  - Taishan People's Hospital, Taishan
  - Taizhou People's Hospital, Taizhou
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Affiliated Hospital of Jiangnan University, Wuxi
  - Wuxi People's Hospital, Wuxi
  - Wuxi Second People's Hospital, Wuxi
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - The People's Hospital of Jiawang District of Xuzhou City, Xuzhou
  - Xuzhou Central Hospital, Xuzhou
  - Yancheng No.1 People's Hospital, Yancheng
  - Affiliated Hospital of Yangzhou University, Yangzhou
  - Subei People's Hospital of Jiangsu province, Yangzhou
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou
  - The 7th People's Hospital of Zhengzhou, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang
  - Zhenjiang First People's Hospital, Zhenjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gulati R, Behfar A, Narula J, Kanwar A, Lerman A, Cooper L, Singh M. Acute Myocardial Infarction in Young Individuals. Mayo Clin Proc. 2020 Jan;95(1):136-156. doi: 10.1016/j.mayocp.2019.05.001. PMID 31902409
- [Background] Bahit MC, Kochar A, Granger CB. Post-Myocardial Infarction Heart Failure. JACC Heart Fail. 2018 Mar;6(3):179-186. doi: 10.1016/j.jchf.2017.09.015. PMID 29496021
- [Background] Heusch G, Libby P, Gersh B, Yellon D, Bohm M, Lopaschuk G, Opie L. Cardiovascular remodelling in coronary artery disease and heart failure. Lancet. 2014 May 31;383(9932):1933-43. doi: 10.1016/S0140-6736(14)60107-0. Epub 2014 May 13. PMID 24831770
- [Background] Juilliere Y, Cambou JP, Bataille V, Mulak G, Galinier M, Gibelin P, Benamer H, Bouvaist H, Meneveau N, Tabone X, Simon T, Danchin N; FAST-MI Investigators. Heart failure in acute myocardial infarction: a comparison between patients with or without heart failure criteria from the FAST-MI registry. Rev Esp Cardiol (Engl Ed). 2012 Apr;65(4):326-33. doi: 10.1016/j.recesp.2011.10.027. Epub 2012 Feb 20. PMID 22357361
- [Background] Bradley EH, Nallamothu BK, Herrin J, Ting HH, Stern AF, Nembhard IM, Yuan CT, Green JC, Kline-Rogers E, Wang Y, Curtis JP, Webster TR, Masoudi FA, Fonarow GC, Brush JE Jr, Krumholz HM. National efforts to improve door-to-balloon time results from the Door-to-Balloon Alliance. J Am Coll Cardiol. 2009 Dec 15;54(25):2423-9. doi: 10.1016/j.jacc.2009.11.003. PMID 20082933
- [Background] Mangin L, Lotfi M, Puie P, Yayehd K, Ispas A, Belle L. [Management of high thrombus burden in primary PCI]. Ann Cardiol Angeiol (Paris). 2017 Dec;66(6):380-384. doi: 10.1016/j.ancard.2017.10.016. Epub 2017 Oct 31. French. PMID 29096903
- [Background] Bai M, Pan CL, Zhao J, Zhao CR, Zhang B, Mu ZY, Meng XX, Zhou XH, Zhu YQ, Zhang Z. [Safety and efficacy of regional transport combined with PCI model in patients with STEMI after thrombolysis in northwest China]. Zhonghua Xin Xue Guan Bing Za Zhi. 2020 Aug 24;48(8):641-647. doi: 10.3760/cma.j.cn112148-20200228-00138. Chinese. PMID 32847319
- [Background] Schwartz R, Weiss AT, Leibowitz D, Rot D, Pollak A, Lotan C, Alcalai R. Thrombolysis followed by coronary angiography versus primary percutaneous coronary intervention in non-anterior ST-elevation myocardial infarction. J Invasive Cardiol. 2013 Dec;25(12):632-6. PMID 24296382
- [Background] Ren K, Gong H, Huang J, Liu Y, Dong Q, He K, Tian L, Zhang F, Yu A, Wu C. Thrombolytic and anticoagulant effects of a recombinant staphylokinase-hirudin fusion protein. Thromb Res. 2021 Dec;208:26-34. doi: 10.1016/j.thromres.2021.10.005. Epub 2021 Oct 14. PMID 34688099
- [Background] Vanderschueren S. [Staphylokinase for a better thrombolytic treatment of heart and platelet diseases]. Verh K Acad Geneeskd Belg. 2000;62(1):69-75. Dutch. PMID 10769618
- [Background] Ueshima S, Matsuo O. Development of new fibrinolytic agents. Curr Pharm Des. 2006;12(7):849-57. doi: 10.2174/138161206776056065. PMID 16515501
- [Background] Yamamoto J, Kawano M, Hashimoto M, Sasaki Y, Yamashita T, Taka T, Watanabe S, Giddings JC. Adjuvant effect of antibodies against von Willebrand Factor, fibrinogen, and fibronectin on staphylokinase-induced thrombolysis as measured using mural thrombi formed in rat mesenteric venules. Thromb Res. 2000 Mar 1;97(5):327-33. doi: 10.1016/s0049-3848(99)00184-x. PMID 10709908
- [Background] Szemraj J, Stankiewicz A, Rozmyslowicz-Szerminska W, Mogielnicki A, Gromotowicz A, Buczko W, Oszajca K, Bartkowiak J, Chabielska E. A new recombinant thrombolytic and antithrombotic agent with higher fibrin affinity - a staphylokinase variant. An in-vivo study. Thromb Haemost. 2007 Jun;97(6):1037-45. doi: 10.1160/th06-10-0562. PMID 17549308
- [Background] Vakili B, Nezafat N, Negahdaripour M, Yari M, Zare B, Ghasemi Y. Staphylokinase Enzyme: An Overview of Structure, Function and Engineered Forms. Curr Pharm Biotechnol. 2017;18(13):1026-1037. doi: 10.2174/1389201019666180209121323. PMID 29424308
- [Background] Li CJ, Huang J, Yang ZJ, Cao KJ. Thrombolytic efficacy of native recombinant staphylokinase on femoral artery thrombus of rabbits. Acta Pharmacol Sin. 2007 Jan;28(1):58-65. doi: 10.1111/j.1745-7254.2007.00455.x. PMID 17184583
- [Background] Nedaeinia R, Faraji H, Javanmard SH, Ferns GA, Ghayour-Mobarhan M, Goli M, Mashkani B, Nedaeinia M, Haghighi MHH, Ranjbar M. Bacterial staphylokinase as a promising third-generation drug in the treatment for vascular occlusion. Mol Biol Rep. 2020 Jan;47(1):819-841. doi: 10.1007/s11033-019-05167-x. Epub 2019 Nov 1. PMID 31677034
- [Background] Vanderschueren S, Barrios L, Kerdsinchai P, Van den Heuvel P, Hermans L, Vrolix M, De Man F, Benit E, Muyldermans L, Collen D, et al. A randomized trial of recombinant staphylokinase versus alteplase for coronary artery patency in acute myocardial infarction. The STAR Trial Group. Circulation. 1995 Oct 15;92(8):2044-9. doi: 10.1161/01.cir.92.8.2044. PMID 7554180
- [Background] Armstrong PW, Burton J, Pakola S, Molhoek PG, Betriu A, Tendera M, Bode C, Adgey AA, Bar F, Vahanian A, Van de Werf F; CAPTORS II Investigators. Collaborative Angiographic Patency Trial Of Recombinant Staphylokinase (CAPTORS II). Am Heart J. 2003 Sep;146(3):484-8. doi: 10.1016/S0002-8703(03)00312-0. PMID 12947367
- See also: Trial Design — https://linkinghub.elsevier.com/retrieve/pii/S0002-8703(23)00168-0